CLINICAL TRIAL: NCT03846050
Title: Risk for Alcohol Impaired Driving: From the Laboratory to the Natural Environment
Brief Title: Alcohol Impaired Driving: From the Laboratory to the Natural Environment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Denis McCarthy, Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 2008051; R01AA019546 (NIH)
Record Dates: First submitted 2019-01-30; First posted 2019-02-19 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Drinking and Driving
Keywords: alcohol impaired driving; decision making; drunk driving; ambulatory assessment
MeSH Terms: conditions — Driving Under the Influence

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to 3 conditions, 2 "active" and one control condition. In the active conditions, participants will receive "warning" messages when their BAC reaches a set threshold that it is not safe for them to drive.
  The two "Active" conditions differ in the timing of their onset of the intervention.
  The control condition will not receive warning and will not report on their driving decision in the moment.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BAC Feedback, immediate onset (Experimental): Participants will receive a"BAC Feedback/Warning" intervention based on their assessed BAC. Participants in this arm will have a warning presented on their smartphone when they provide a breath sample that indicated their BAC has reached a set limit. The cutpoint for this warning is not disclosed but is well below the legal limit for driving. Warning will notify them that their results indicate it is not safe for them to drive.
  In this condition, participants will start their 6 week AA portion of their participation immediately after their laboratory session, and will be followed for 6 weeks afterwards.
  Comparisons between the two experimental conditions will allow for inferences about the onset and offset of any effects of the "BAC Feedback/Warning" intervention.
  Interventions: Behavioral: BAC feedback/warning
- BAC Feedback, delayed onset (Experimental): Participants will receive the "BAC Feedback/Warning" intervention based on their assessed BAC during drinking events.The cutpoint for this warning is not disclosed but is well below the legal limit for driving. Warning will notify them that their results indicate it is not safe for them to drive.
  In this condition, participants will be followed for 6 weeks after their laboratory session prior to starting their 6 week AA portion of their participation.
  Comparisons between the two experimental conditions will allow for inferences about the onset and offset of any effects of the "BAC Feedback/Warning" intervention.
  Interventions: Behavioral: BAC feedback/warning
- Minimal Assessment Control (Placebo Comparator): Participants will receive the "No BAC Feedback/Warning" intervention. Participants in this condition will complete the laboratory and interview portions of the project. However the AA portion of the project will not contain warning about their BAC (No BAC Feedback/Warning) and will ask fewer questions regarding their AID decisions.
  The role of this condition is to provide a baseline comparison of AID behavior for the two active assessment conditions.
  Interventions: Behavioral: No BAC feedback/warning

INTERVENTIONS:
Behavioral: BAC feedback/warning — Participants will receive a warning when their BAC reaches a set limit. The cutpoint for this warning is not disclosed but is well below the legal limit for driving. Warning will notify them that their results indicate it is not safe for them to drive.
  Arms: BAC Feedback, delayed onset; BAC Feedback, immediate onset
Behavioral: No BAC feedback/warning — Participants will receive no information on their current intoxication and will be asked to report less information on their driving decisions.
  Arms: Minimal Assessment Control

SUMMARY:
This project combined laboratory and ambulatory assessment (AA) methods to test decision making associated with alcohol impaired driving (AID). Participants will complete a laboratory alcohol administration session followed by 6 weeks of mobile assessment. Data from drinking events will be examined to test how individuals make choices about driving or not after consuming alcohol.

DETAILED DESCRIPTION:
Building on laboratory findings from the the PI's (McCarthy) previous work, this project is designed to test AID decision making in both the lab and the natural drinking environment in which AID decisions are made.

Participants complete a laboratory alcohol administration session followed by six weeks of multi-method ambulatory assessment. The ambulatory assessment component will include participant report via smartphone, portable breathalizer (BACtrack), and location and movement data passively collected by the smartphone GPS/accelerometer. The combination of these methods will allow for the integration of subjective (e.g., perceived intoxication) and objective (e.g., BrAC, calculated drinking location) data for each drinking episode.

Aim 1 of the project is to test laboratory measures as prospective predictors of AID and examine the role of event-level influences on specific AID decisions.

Aim 2 of the proposed project is to test the potential for a novel intervention to reduce AID using mobile technology. Participants will be randomly assigned to either a full ambulatory assessment or a minimal assessment control condition. The timing of the introduction of AA will also be manipulated within the full ambulatory assessment condition. This design will allow us to test whether the introduction of ambulatory assessment produces changes in AID behavior, as well as whether such changes persist once ambulatory assessment is discontinued. Changes made to the revised application are aimed at ensuring the achievement of both study aims. If Aim 2 is achieved and ambulatory assessment alters AID behavior, the combination of the minimal assessment control condition and the full assessment condition prior to the introduction of ambulatory assessment has sufficient sample size and power to test Aim 1 hypotheses.

ELIGIBILITY:
Inclusion Criteria:

* moderate to heavy drinkers must drive regularly report recent binge drinking fluent in english

Exclusion Criteria:

* not in treatment for substance use disorder or other psychiatric disorders BMI under 30 no medical conditions contraindicating alcohol consumption

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 230 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Alcohol impaired driving behavior | 12 weeks
  Participants will provide self-reported driving behavior (yes/no driven a vehicle) after drinking alcohol during the AA portion. This assessment will be taken from their daily smartphone responses.
Alcohol impaired driving behavior (retrospective) | 12 weeks
  Participants will provide self-reported driving behavior (yes/no driven a vehicle) after drinking alcohol retrospectively during interview sessions. Participants will complete regular phone interview where their daily driving and drinking behavior will be assessed. The outcome measure of interest will be days when participants report driving (yes/no) after consuming alcohol.
Alcohol impaired driving intentions | 6 weeks
  Participants will provide self-reported intentions to drive after drinking alcohol (Would you drive now? Yes/no) from daily assessments during the AA portion of the project.

SECONDARY OUTCOMES:
Perceived risk of driving | 6 weeks
  Participants will report their perceived risk of driving (1 to 4 scale, "Not Dangerous to Very Dangerous") given their current level of impairment during AA portion of project.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haney AM, Motschman CA, Warner OM, Wesley RL, Wycoff AM, Trull TJ, McCarthy DM. Comparing associations between mood and breath alcohol concentration in the laboratory and natural environment. Psychol Addict Behav. 2022 Nov;36(7):885-894. doi: 10.1037/adb0000814. Epub 2022 Feb 7. PMID 35129995